CLINICAL TRIAL: NCT00004908
Title: Autologous Blood Stem Cell Transplantation in Patients With Hodgkin's Disease and Non-Hodgkin's Lymphoma With High-Dose Cyclophosphamide, Total Body Irradiation and Involved-Field Radiation Therapy
Brief Title: Radiation Therapy and Cyclophosphamide Plus Peripheral Stem Cell Transplantation in Treating Patients With Recurrent or Refractory Hodgkin's Disease or Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NU 87H5T; NU-87H5T; NCI-G00-1693
Record Dates: First submitted 2000-03-07; First posted 2004-03-03 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent childhood large cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cyclophosphamide
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage cancer cells. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Peripheral stem cell transplantation may allow doctors to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of radiation therapy and cyclophosphamide plus peripheral stem cell transplantation in treating patients who have recurrent or refractory Hodgkin's disease or non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity of autologous peripheral blood stem cell transplantation following involved field radiotherapy, high dose cyclophosphamide, and total body irradiation in patients with recurrent or refractory Hodgkin's disease or non-Hodgkin's lymphoma. II. Determine the response in patients treated with this regimen.

OUTLINE: Patients undergo involved field radiotherapy on days -16 to -7. Patients receive cyclophosphamide IV over 2 hours on days -6 and -5. Patients undergo total body irradiation twice daily on days -4 to -1. Autologous peripheral blood stem cells are reinfused on day 0. Patients are followed every month for 1 year.

PROJECTED ACCRUAL: Not specified

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven Hodgkin's disease or non-Hodgkin's lymphoma that is refractory to standard therapy or has relapsed following initial response Eligible non-Hodgkin's lymphoma: Low grade Intermediate grade Immunoblastic large cell lymphoma (high grade) Eligible for involved field radiotherapy, cyclophosphamide, and total body irradiation No CNS non-Hodgkin's lymphoma or Hodgkin's disease A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: Physiologic age 65 and under Performance status: ECOG 0-2 Life expectancy: At least 2 months Hematopoietic: Not specified Hepatic: Not specified Renal: Creatinine less than 1.5 mg/dL OR Creatinine clearance greater than 50 mL/min if creatinine 1.5-2 mg/dL Cardiovascular: No active heart disease (congestive heart failure, history of myocardial infarction within the past 3 months, or significant arrhythmia) requiring medication Pulmonary: No nonneoplastic pulmonary disease (e.g., chronic obstructive pulmonary disease) that would preclude intensive chemotherapy DLCO at least 50% predicted* FEV1 and/or FVC at least 75% predicted* * Unless due to underlying lymphoma or Hodgkin's disease Other: No other concurrent medical condition that would preclude aggressive cytotoxic chemotherapy HIV negative No clinical evidence of AIDS

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-11; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane N. Winter, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States